CLINICAL TRIAL: NCT01452295
Title: Registry Protocol for Tracking the Incidence of Transplant, the Incidence and Type of Cancer, and Survival Rate of Subjects Participating in Protocol VTI-206 (NCT00973817)
Brief Title: Registry Protocol for Tracking Trial Subjects After VTI-206 Study Completion
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Subjects from lead-in study VTI-206 - NCT00973817 lost to follow-up before enrollment in VTI-207 (NCT1452295)
Sponsor: Vital Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: VTI-207
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Acute Liver Failure
Keywords: liver; liver failure; acute liver failure; ELAD; alcoholic hepatitis; acute on chronic hepatitis
MeSH Terms: conditions — Liver Failure, Acute; Liver Failure; Hepatitis, Alcoholic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AOCH patients (Experimental): Patients with acute on chronic hepatitis
  Interventions: Drug: ELAD (Extracorporeal Liver Assist System)
- AAH patients (Experimental): Patients with acute alcoholic hepatitis
  Interventions: Drug: ELAD (Extracorporeal Liver Assist System)

INTERVENTIONS:
Drug: ELAD (Extracorporeal Liver Assist System) — ELAD (Extracorporeal Liver Assist System)

SUMMARY:
VTI-207 (NCT01452295) is designed to follow subjects, both treated and control, for five years after their completion of study participation in protocol VTI-206 (NCT00973817) to gather information relating to the incidence of liver transplant, the incidence and type of cancer (if any), and survival.

DETAILED DESCRIPTION:
Vital Therapies, Inc. (VTI) is conducting clinical trial VTI-206 in which subjects with acute on chronic hepatitis (AOCH) and acute alcoholic hepatitis (AAH) are treated with the ELAD system to assess the safety and efficacy of this therapy. The ELAD system incorporates cloned immortalized human liver cells (C3A cells). A hypothetical risk exists that, over an extended period of time, there may be an increased incidence of tumor in subjects treated with ELAD.

The company is also collecting data related to whether a patient received a liver transplant and on survival.

ELIGIBILITY:
Inclusion Criteria:

* Subjects participating in the VTI-206 clinical trial.

Exclusion Criteria:

* Subjects not participating in the VTI-206 clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Gather data | Five years post study participation
  See previous description

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Ashley, Study Director — Vital Therapies, Inc.